CLINICAL TRIAL: NCT01150370
Title: A Pivotal Study to Assess the Safety and Efficacy of The PrePex System, a Male Circumcision Device and Methodology for Rapid Scale up of Painless and Bloodless National Circumcision Programs, in Urban and Remote Rural Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Health, Rwanda (Other Government)
Collaborators: Ministry of Defence, Rwanda (Unknown)
Responsible Party: Ministry of Health, Rwanda, Ministry of Health, Rwanda
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CMT-01
Record Dates: First submitted 2010-06-23; First posted 2010-06-25 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2010-12

CONDITIONS: Male Circumcision; HIV Prevention; HIV Infections
Keywords: male circumcision; HIV; Rwanda; HIV Seronegativity
MeSH Terms: conditions — HIV Infections

ARMS (1):
- Males undergoing circumcision (Experimental)
  Interventions: Device: The PrePex a novel device for adult male circumcision

INTERVENTIONS:
Device: The PrePex a novel device for adult male circumcision — The PrePex System was designed to enable safe, effective, painless and bloodless male circumcision programs. The PrePex System includes a simple, disposable device that is easy to use and can be deployed by minimally trained healthcare professionals, without the need for sterile, hospital settings.

SUMMARY:
The protocol, approved by the Rwanda National Ethical Committee, was issued to assess the safety and efficacy of the circumcision device for applying it to the national scale up of adult male circumcision in Rwanda

DETAILED DESCRIPTION:
Multiple randomized and controlled studies (WHO, USAID, UNAIDS) have proven that circumcised men in high risk areas reduce their risk of HIV infection by 60%.

The Government of Rwanda has ranked HIV prevention as a top priority item, and wishes to decrease the HIV incidence in the country by 50%. As part of a holistic HIV prevention approach, we decided to embark upon a process of national scale up of adult male circumcision. The national HIV prevention plan calls for voluntary MC of 2 million adults by the end of 2012.

The PrePex System was designed to enable safe, effective, painless and bloodless male circumcision programs, to support global public health efforts to stop the spread of HIV.

The PrePex System includes a simple, disposable device that is easy to use and can be deployed by minimally trained healthcare professionals, in urban or rural settings, without the need for sterile, hospital settings. As such, The PrePex System places minimal burden on the existing health care infrastructure to accomplish national circumcision programs.

The protocol, approved by the Rwanda National Ethical Committee, was issued to assess the safety and efficacy of the circumcision device for applying it to the national scale up of adult male circumcision in Rwanda.

ELIGIBILITY:
Inclusion Criteria:

* Male of ages 18 - 54 years
* Subject wants to be circumcised
* Uncircumcised
* HIV sero-negative Agrees to undergo measurements of width of the penis at different areas in flaccid status
* Able to understand the study procedures and requirements
* Agrees to abstain sexual intercourse and to keep caution not directly rub the cut area if masturbating, until the end of the follow-up that may take up to 6 weeks
* Subject able to comprehend and freely give informed consent for participation in this study and is considered by the investigator to have good compliance for the study

Exclusion Criteria:

* Active genital infection, anatomic abnormality or other condition, which in the opinion of the investigator prevents the subject from undergoing a circumcision
* HIV sero-positive
* Subject with the following diseases: phimosis, paraphimosis, warts under the prepuce, torn or tight frenulum, narrow prepuce, hypospadias
* Diabetes mellitus
* Subject who have an abnormal penile anatomy or any penile diseases
* Subject that to the opinion of the investigator is not a good candidate

Ages: 18 Years to 54 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The efficacy and safety of The PrePex System for adult male circumcision in Rwanda | 4 week post-procedure follow up appointment and examination
  Outcome measures will include:
  Number of Participants with Adverse Events as a Measure of Safety,
  Pain as measured by Visual Analogue Scale (VAS),
  Wound healing rate.

SECONDARY OUTCOMES:
Operational scalability to mass scale up program | four week post-procedure follow up appointment and examination
  Outome measure include:
  Duration required by diffrent personnel to perform the procedure Procedure performance by nurses
satisfaction & acceptability of patients | 4 weeks follow up
  Outcome measure include:
  Quality of life and satisfaction questionnaire
Guidelines for utility in scale up mass circumcision program | 4 weeks follow up
  Outcome measure includes:
  Physicians questionnaire on the clinical and practical performance of the procedure
compliance with post procedure instructions | 4 weeks follow up
  Outcome measure include:
  Weekly follow up visits post procedure, compliance with post procedure instructions questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Jean Paul Bitega, M.D., Principal Investigator — Kanombe Military Hospital
Locations (1):
- Kanombe Military Hospital, Kigali, Kigali, Rwanda

REFERENCES:
- See also: Related Info — http://www.moh.gov.rw